CLINICAL TRIAL: NCT04795726
Title: A Clinical Trial Collecting Data From Routine Ophthalmological Examinations of Patients Who Were Randomized to Either Finerenone or Placebo in the Two Bayer-sponsored Phase 3 Clinical Trials FIDELIO-DKD and FIGARO-DKD to Investigate the Effect of Finerenone on Delaying the Progression of Diabetic Retinopathy
Brief Title: A Study That Uses Data From Routine Eye Examinations of Patients Participating in Studies FIDELIO-DKD and FIGARO-DKD to Explore Whether Finerenone Can Delay the Progression of a Diabetes Complication That Affects the Eyes (Diabetic Retinopathy, DR)
Acronym: DeFineDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 21618; 2020-003865-20 (EudraCT Number)
Record Dates: First submitted 2021-02-26; First posted 2021-03-12 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients received treatment in phase 3 clinical trials FIDELIO-DKD (16244) and FIGARO-DKD (17530).
  Interventions: Drug: Finerenone (BAY94-8862)
- Placebo group (Placebo Comparator): Patients received placebo in phase 3 clinical trials FIDELIO-DKD (16244) and FIGARO-DKD (17530).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone (BAY94-8862) — 10 mg or 20 mg Finerenone tablet to be given orally, once daily, administered in the FIDELIO-DKD or FIGARO-DKD clinical trial.
  Arms: Treatment group
Drug: Placebo — Matching placebo to be taken orally, once daily, administered in the FIDELIO-DKD or FIGARO-DKD clinical trial.
  Arms: Placebo group

SUMMARY:
Diabetic retinopathy (DR) is a diabetes complication caused by damage to the small blood vessels inside the retina at the back of the eye. Diabetic retinopathy may cause mild vision problems or eventually blindness. Diabetes is a condition that makes your blood sugar levels higher than they should be.

In the early stages of diabetic retinopathy - called non-proliferative diabetic retinopathy (NPDR)- increased blood sugar levels lead to damage to the tiny blood vessels of the retina. This damage results in small outpouchings of the vessel lumens leading to rupture. At the same time the blood vessels can leak and making the retina swell and can cause so called macula edema. In these early stages of DR current treatment to reduce the risk of this eye complication is focused on controlling blood sugar levels and blood pressure.

Participants in this study have NPDR, Type 2 Diabetes (T2D) and Chronic Kidney Disease (CKD), a condition in which the kidneys become damaged and do not work as they should. These participants are already taking part in one of the phase 3 studies (FIDELIO-DKD and FIGARO-DKD). They study the effect of Finerenone on delaying kidney disease progression and reducing the risk of events that may cause damage to the heart and blood vessels To learn more about the effect of Finerenone on diabetic retinopathy, data from routine eye examinations performed during the two phase 3 studies will be collected and analyzed. All male and female participants included in this study are at least 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in DeFineDR
* Included in FIDELIO-DKD or FIGARO-DKD, and with DR as medical history
* Documented NPDR in at least one eye, as documented by ophthalmological records within 6 months prior to baseline in FIDELIO-DKD or FIGARO-DKD, and up to one month after baseline in FIDELIO-DKD or FIGARO-DKD
* An ophthalmological assessment available 6 month before or maximum 1 month after the baseline examination in FIDELIO-DKD or FIGARO-DKD, and at least one additional assessment afterwards.

Exclusion Criteria:

* Participants with PDR, macular edema or anterior segment complications present at baseline in FIDELIO-DKD or FIGARO-DKD in at least one eye.
* Participants with any documentation of prior or planned retinal laser treatment, intravitreal injection or vitrectomy at baseline in FIDELIO-DKD or FIGARO-DKD in at least one eye.
* Participants with any other retinal disease documented at baseline in FIDELIO-DKD or FIGARO-DKD in at least one eye that would likely interfere with the study objectives (e.g. neovascular age-related macular degeneration or retinal vein occlusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with progression of non-proliferative diabetic retinopathy (NPDR) | After start of treatment until end of Year 2
  Progression of non-proliferative diabetic retinopathy (NPDR) defined by the occurrence of vision-threatening events i.e. proliferative diabetic retinopathy (PDR), diabetic macular edema (DME), anterior segment neovascularization (ASN) until the end of Year 2 after start of treatment

SECONDARY OUTCOMES:
Proportion of participants with progression of non-proliferative diabetic retinopathy (NPDR) | After start of treatment until end of Year 1
  Progression of non-proliferative diabetic retinopathy (NPDR) defined by the occurrence of vision-threatening events i.e. proliferative diabetic retinopathy (PDR), diabetic macular edema (DME), anterior segment neovascularization (ASN) until the end of Year 1 after start of treatment
Proportion of participants with progression of NPDR to Proliferative Diabetic Retinopathy (PDR) | After start of treatment until end of Year 1, and until the end of Year 2
Proportion of participants with diabetic macular edema (DME) | After start of treatment until end of Year 1 and end of Year 2
Proportion of participants with anterior segment neovascularization (ASN) | After start of treatment until end of Year 1 and end of Year 2
Change in severity of diabetic retinopathy (DR) | From strat of treatment to the end of Year 1 and end of Year 2
  Severity grade of DR:
  No DR NPDR (mild or moderate) NPDR (severe) PDR

CONTACTS AND LOCATIONS:
Locations (11):
- Bulgaria (7):
  - Med Centre Diamedical 2013, Dimitrovgrad
  - MHAT Sveta Karidad, Plovdiv
  - MHAT Hadzhi Dimitar, Sliven
  - MHAT Dr. Bratan Shukerov AD, Smolyan
  - DCC Aleksandrovska, Sofia
  - MCOMH Preventsia-2000, Stara Zagora
  - MHAT Sveti Pantaleymon - Yambol, Yambol
- United Kingdom (4):
  - Southmead Hospital, Bristol, Avon
  - St Richard's Hospital, Chichester, West Sussex
  - Royal London Hospital, London
  - King's College Hospital - NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/